CLINICAL TRIAL: NCT02061306
Title: Celiac Disease Genomic Environmental Microbiome and Metabolomic (CDGEMM) Study
Brief Title: Celiac Disease Genomic Environmental Microbiome and Metabolomic Study
Acronym: CDGEMM
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Roma La Sapienza (Other); Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Alessio Fasano, Chief of Pediatric Gastroenterology and Nutrition, Massachusetts General Hospital
Other Study IDs: 2013P001965
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Celiac Disease
Keywords: Celiac disease; coeliac disease; microbiome; gluten; infants; pregnancy; genetic
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Periodic stool and blood collection from infant, optional cord blood sample. Optional collection of maternal stool samples prenatal and enrollment, including enrollment breast milk sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with a first-degree relative with celiac disease: Infants who have a first-degree relative diagnosed with celiac disease.

SUMMARY:
Celiac disease (CD) is a complex disease caused by eating gluten, a protein contained in wheat, rye, and barley. It is well known that many factors contribute to the development of CD, including the genes that you have and the foods that you eat. In the CDGEMM study, we will consider as many of these factors as possible and study how they each contribute to disease development. If the investigators find that any one factor, or combination of factors, increases the risk of developing CD, we will be able to apply this information and help prevent or detect disease in high-risk children in the future.

DETAILED DESCRIPTION:
The CDGEMM study will address genomic, environmental, microbiome, and metabolomic factors that could affect the development of CD.

Genomic: The investigators will study children who have a first degree relative with celiac disease so that we can understand how their genes may contribute to whether they develop CD or not. Scientists and doctors are already aware of one group of genes, called the HLA DQ2 and DQ8 genes, which are involved in the development of CD. These genes are necessary for development of CD, but cannot alone predict who will develop the disease. The investigators hope that the CDGEMM study will help to not only learn more about these specific genes, but also identify other genes that could make it easier to predict who will develop CD.

Environmental: When infants enroll, the investigators will record information about their environment including whether they were born vaginally or by Cesarean section and whether they were given antibiotics. Over time, the investigators will also consider other parts of the infant's medical history including feeding modality (breastfeeding versus formula feeding), illnesses, infections, and growth to understand if any of this information is related to CD development. Since the investigators will follow infants until they reach 5 years of age, the investigators will update this information every six months to understand how changes might affect if the child develops CD or not.

Microbiome: Our gut, compromised of the small and large intestine, contains many types of bacteria. These bacteria that live in the gut normally help to break down and digest food, provide our bodies with energy, and make vitamins that our bodies need. This diverse community of bacteria is called the gut microbiome. A main goal of the CDGEMM study is to understand how the microbiome is affected by other factors, like foods or antibiotic drugs, and how this may affect the development of CD. It is possible that learning about the types of bacteria living in the gut before and after disease development may help us predict who will develop CD before it happens.

Metabolomic: The processes that occur in our gut, such as the digestion of foods and production of vitamins, create products that are called metabolites. The specific metabolites that we produce differ from person to person and depend on many factors, including the genes that we have, the members of the gut microbiome, and the foods that we eat. We will study the infant's unique metabolomic profile (metabolites that the infant produces) to understand if there is a specific profile associated with CD.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and infants less than 6 months of age who have not been introduced to solid foods (exclusive breast milk or formula diet)
* First-degree relatives of patients affected with biopsy-proven CD

Exclusion Criteria:

* Infants older than 6 months of age
* Inability or unwillingness of legal guardian/representative to give written informed consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns and infants younger than 6 months who are first-degree relatives of CD patients (at least one parent or sibling affected with biopsy-proven CD) are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in composition of the microbiota of CD in at-risk infants using culture-independent high-throughput sequence analysis of the 16S rRNA genes using the Illumina sequencing platform. | Every six months through five years of age with specific focus on time of gluten introduction, time at which gluten tolerance is lost and autoimmunity develops (if applicable), and parallel time points in infants who do not go on to develop autoimmunity
  We will use stool samples collected over time to survey the microbial community in order to establish microbiota patterns associated with CD autoimmunity.

SECONDARY OUTCOMES:
Change in gut permeability measured by serum zonulin levels and loss of gluten tolerance measured by increased expression of pro-inflammatory cytokines and appearance of anti-tTg antibodies. | Every six months until age 3. Every year thereafter until age 5.
  We anticipate that timing of gluten introduction in the infant's diet will influence shift in enterotype and metatranscriptome profile with subsequent increase in gut permeability and loss of gluten tolerance.

OTHER OUTCOMES:
Comparison of the characterization of infants' metabotypes (metabolomes) using an established and proven commercial metabolomics technology platform by Metabolon, Inc. | Every six months through five years of age with specific focus on time of gluten introduction, time at which gluten tolerance is lost and autoimmunity develops (if applicable), and parallel time points in infants who do not go on to develop autoimmunity
  Our preliminary data suggest that individual metabolomic phenotypes (which are a result of gene-diet-gut microbiome interactions) can help define specific enterotypes associated to loss of gluten tolerance in infants genetically at risk of CD.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Fasano, MD, Principal Investigator — Massachusetts General Hospital; Maureen M. Leonard, MD, Study Chair — Massachusetts General Hospital
Locations (2):
- MassGeneral Hospital for Children, Boston, Massachusetts, United States
- University of Roma La Sapienza, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leonard MM, Karathia H, Pujolassos M, Troisi J, Valitutti F, Subramanian P, Camhi S, Kenyon V, Colucci A, Serena G, Cucchiara S, Montuori M, Malamisura B, Francavilla R, Elli L, Fanelli B, Colwell R, Hasan N, Zomorrodi AR, Fasano A; CD-GEMM Team. Multi-omics analysis reveals the influence of genetic and environmental risk factors on developing gut microbiota in infants at risk of celiac disease. Microbiome. 2020 Sep 11;8(1):130. doi: 10.1186/s40168-020-00906-w. PMID 32917289
- See also: CDGEMM Study Website — http://www.CDGEMM.org